CLINICAL TRIAL: NCT01398410
Title: Long-term Prevention of Recurrent Gastric or Duodenal Ulcers Caused by Low-dose Aspirin With Rabeprazole (E3810) Treatment. - A Multicenter, Randomized, Parallel-group, Open-label Trial-
Brief Title: Long-term Prevention of Recurrent Gastric or Duodenal Ulcers Caused by Low-dose Aspirin With Rabeprazole (E3810) Treatment (Planetarium Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E3810-J081-309
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Gastric Ulcers Duodenal Ulcers Caused by Low-dose Aspirin
Keywords: Rabeprazole; proton pump inhibitor; Acetylsalicylic Acid; Aspirin; Gastric Ulcer; Duodenal Ulcer
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — Rabeprazole

ARMS (2):
- Rabeprazole 5 mg (Experimental)
  Interventions: Drug: Rabeprazole
- Rabeprazole 10 mg (Experimental)
  Interventions: Drug: Rabeprazole

INTERVENTIONS:
Drug: Rabeprazole — Participants received rabeprazole 5 mg tablets and rabeprazole 10 mg matched placebo tablets orally, once daily
  Other Names: E3810, Pariet/Aciphex
  Arms: Rabeprazole 5 mg
Drug: Rabeprazole — Participants received rabeprazole 10 mg tablets and rabeprazole 5 mg matched placebo tablets orally, once daily
  Other Names: E3810, Pariet/Aciphex
  Arms: Rabeprazole 10 mg

SUMMARY:
The primary objective of this study to examine the long-term safety of rabeprazole 5 mg or 10 mg tablets administered once daily in participants who were confirmed to have no recurrence of gastric or duodenal ulcer by endoscopic examination at the end of 24 weeks of treatment in the E3810-J081-308 (NCI01397448) [Double-Blind Phase] study. From a total of 420 participants who completed the E3810-J081-308 study, 328 entered the E3810-J081-309 (NCT01398410) study.

DETAILED DESCRIPTION:
The E3810-J081-309 consisted of two arms: the long-term rabeprazole groups (participants from the rabeprazole 5 or 10 mg arm of the E3810-J081-308 study who entered the rabeprazole 5 mg or 10 mg arm of the E3810-J081-309 study) and the newly-initiated rabeprazole groups (participants from the teprenone 150 mg arm of the E3810-J081-308 study who entered the rabeprazole 5 mg or 10 mg arm of the E3810-J081-309 study).

ELIGIBILITY:
Inclusion Criteria

* Confirmed to have no recurrence of gastric or duodenal ulcer by endoscopy at the end of 24 weeks of treatment in study E3810-J081-308.
* Need to continue receiving low-dose aspirin (81 mg/day or 100 mg/day) during this study.

Exclusion Criteria

-Confirmed to have a recurrence of gastric or duodenal ulcer at the end of 24 weeks of treatment in study E3810-J081-308 (at the start of this trial) and thus are withdrawn from the trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sugisaki, Study Director — Japan/Asia Clinical Research Product Creation Unit
Locations (50):
- Japan (50):
  - Kasugai, Aichi-ken
  - Nagoya, Aichi-ken
  - Ichikawa, Chiba
  - Chikushino-shi, Fukuoka
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Gifu, Gifu
  - Maebashi, Gunma
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Tomakomai, Hokkaido
  - Itami, Hyōgo
  - Kobe, Hyōgo
  - Hitachi, Ibaraki
  - Fujisawa, Kanagawa
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Kitakyushu, Kitakyushu
  - Kochi, Kochi
  - Hitoyoshi, Kumamoto
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Ebino, Miyazaki
  - Miyazaki, Miyazaki
  - Chikuma, Nagano
  - Matsumoto, Nagano
  - Nagano, Nagano
  - Suzaka, Nagano
  - Nagasaki, Nagasaki
  - Beppu, Oita Prefecture
  - Ōita, Oita Prefecture
  - Yufu, Oita Prefecture
  - Daitō, Osaka
  - Hirakat, Osaka
  - Matsubara, Osaka
  - Osaka, Osaka
  - Takatsuki, Osaka
  - Yao, Osaka
  - Karatsu, Saga-ken
  - Saga, Saga-ken
  - Ureshino, Saga-ken
  - Izumo, Shimane
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Ohtawara, Tochigi
  - Mitaka, Tokyo
  - Setagaya City, Tokyo
  - Shinjuku, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From a total of 420 participants who completed the E3810-J081-308 (NCT01397448) study, 405 entered the E3810-J081-309 (NCT01398410) study.
Groups:
- Rabeprazole 5 mg: Participants received rabeprazole 5 mg tablets and rabeprazole 10 mg matched placebo tablets orally, once daily
- Rabeprazole 10 mg: Participants received rabeprazole 10 mg tablets and rabeprazole 5 mg matched placebo tablets orally, once daily
Period: Overall Study
Arm/Group | Rabeprazole 5 mg | Rabeprazole 10 mg
Started | 201 (Treated participants (all participants who received at least one dose of rabeprazole).) | 204
Completed | 143 | 148
Not Completed | 58 | 56
Not completed — Adverse Event | 12 | 16
Not completed — Participants Choice | 8 | 11
Not completed — Inadequate Therapeutic Effect | 2 | 0
Not completed — Other | 36 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabeprazole 5 mg | Rabeprazole 10 mg | Total
Number analyzed (Participants) | 201 | 204 | 405
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.4 (8.5) | 70.1 (9.3) | 69.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 153 | 152 | 305

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered with the study drug. A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening (ie, the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was as a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). In this study, treatment emergent AEs (defined as an AE (serious/non-serious) that started/increased in severity on/after the first dose of study drug up to 30 days after the final dose of study drug) were assessed. The data is presented as percentage of participants with treatment emergent AEs.
Time Frame: For each participant, from administration of first dose of study drug (rabeprazole) up to 30 days from administration of last dose of study drug (rabeprazole) or up to 76 weeks (including data from the Double-Blind Phase)
Population: The analysis was performed using Safety Analysis Set, defined as all participants who received at least one dose of rabeprazole.
Measure: Number; unit: Percentage of participants
Arm/Group | Rabeprazole 5 mg | Rabeprazole 10 mg
Number analyzed (Participants) | 201 | 204
Percentage of participants | 77.1 | 83.8

2. Secondary Outcome: Cumulative Recurrent Rate of Gastric or Duodenal Ulcers
Description: Mucosal injuries with a white coat measuring greater than or equal to 3 mm in diameter was diagnosed as ulcers. When ulcer was confirmed by endoscopic examination during the trial, it was regarded as recurrence of ulcer and the trial was discontinued for the participant involved. The presence or absence of ulcer recurrence was determined by the endoscopy central review panel that were blinded to the investigators' assessments. Cumulative recurrent rate was estimated by the Kaplan-Meier method. The data is presented as percentage of participants with cumulative recurrent rate of gastric or duodenal ulcers.
Time Frame: Baseline, Week 12, Week 24, Week 52, and Week 76 (including data from the Double-Blind Phase)
Population: The analysis was performed using Full Analysis Set, defined as all participants who received at least one dose of rabeprazole, with at least one post-initiation endoscopic assessment results, and showed no ulcers on baseline endoscopy; excluding participants from the newly-initiated rabeprazole groups of study E3810-J081-309.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rabeprazole 5 mg | Rabeprazole 10 mg
Number analyzed (Participants) | 150 | 151
Percentage of participants
  Baseline (N=150, 151) | 0 [0 to 0] | 0 [0 to 0]
  Week 12 (N=150, 151) | 1.3 [0.34 to 5.23] | 0 [0 to 0]
  Week 24 (N=139, 142) | 2.8 [1.04 to 7.17] | 1.4 [0.35 to 5.51]
  Week 52 (N=107, 121) | 3.7 [1.53 to 8.64] | 2.2 [0.72 to 6.75]
  Week 76 (N=93, 96) | 3.7 [1.53 to 8.64] | 2.2 [0.72 to 6.75]

ADVERSE EVENTS:
Time Frame: For each participant, from administration of first dose of study drug (rabeprazole) up to 30 days from administration of last dose of study drug or up to 76 weeks (including data from the Double-Blind Phase)
Description: In this study, treatment emergent AEs (defined as an AE (serious/non-serious) that started/increased in severity on/after the first dose of study drug (rabeprazole) up to 30 days after the final dose of study drug) were assessed.
Groups:
- Rabeprazole10 mg: Participants received rabeprazole 10 mg tablets and rabeprazole 5 mg matched placebo tablets orally, once daily
Arm/Group | Rabeprazole 5 mg | Rabeprazole10 mg
Serious Adverse Events (participants affected / at risk) | 33/201 | 30/204
Other Adverse Events (participants affected / at risk) | 89/201 | 99/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole 5 mg (N=201) | Rabeprazole10 mg (N=204)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 3 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 1 | 0
Artery dissection (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole 5 mg (N=201) | Rabeprazole10 mg (N=204)
Diarrhoea (Gastrointestinal disorders) | 11 | 16
Constipation (Gastrointestinal disorders) | 9 | 16
Nasopharyngitis (Infections and infestations) | 64 | 57
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 13
Contusion (Injury, poisoning and procedural complications) | 13 | 7
Eczema (Skin and subcutaneous tissue disorders) | 6 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other